CLINICAL TRIAL: NCT02281500
Title: Multicenter, Prospective, Open-Label, Single-Arm Trial to Evaluate the Pharmacokinetics, Efficacy, and Safety of Human Plasma-Derived Fibrinogen (FIB Grifols) in Patients With Congenital Afibrinogenemia
Brief Title: Pharmacokinetics, Efficacy, and Safety of Human Plasma-Derived Fibrinogen (FIB Grifols) in Participants With Congenital Afibrinogenemia
Acronym: IG0902
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Collaborators: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG0902
Record Dates: First submitted 2014-10-24; First posted 2014-11-03 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Congenital Afibrinogenemia
MeSH Terms: conditions — Afibrinogenemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single (Experimental): Human Plasma-Derived Fibrinogen Concentrate Grifols (FIB Grifols)
  Interventions: Biological: Human Plasma-Derived Fibrinogen Concentrate

INTERVENTIONS:
Biological: Human Plasma-Derived Fibrinogen Concentrate — A sterile freeze-dried fibrinogen concentrate filled in vials containing 1 g of FIB Grifols. FIB Grifols contains 20 mg/ml of active substance fibrinogen when reconstituted.
  Other Names: FIB Grifols

SUMMARY:
The main objective of this study was to evaluate the pharmacokinetics (PK), efficacy, and safety of human plasma-derived fibrinogen concentrate FIB Grifols after a single-dose 70 milligrams/kilogram (mg/kg) body weight administration.

DETAILED DESCRIPTION:
This study is a phase I-II, multi-center, prospective, open-label, single-arm, clinical trial to evaluate Pharmacokinetic (PK), efficacy, and safety of human plasma-derived fibrinogen concentrate (FIB Grifols) in adult and pediatric participants with congenital afibrinogenemia.

Approximately 10 adult participants (≥18 years) with congenital afibrinogenemia will be administered a single dose of FIB Grifols at 70 mg/kg body weight and will be followed for PK, efficacy, and safety assessments.

After the safety of fibrinogen concentrate FIB Grifols is assessed in at least 10 adult participants and no safety issues are raised by the sponsor, the study will start to enroll approximately 10 pediatric subjects (<18 years) who will be dosed with study drug and followed for PK, efficacy, and safety assessments.

All enrolled participants (both adult and pediatric) will have documented congenital fibrinogen deficiency manifested as afibrinogenemia but will not have received any fibrinogen-containing product therapy within the preceding 21 days before the infusion of study drug.

All participants (both adult and pediatrics) will be infused with the investigational product at 70 mg/kg body weight. PK parameters that will be calculated from plasma fibrinogen levels measured at different time points include: incremental in vivo recovery [IVR], area under the curve (AUC) calculated as AUC from zero to 14 days (AUC^0-14days) and AUC from zero to infinity (AUC^0-∞), maximum plasma concentration (C^max), time to the observed maximum plasma concentration (t^max), half-life (t^1/2), mean residence time (MRT), volume of distribution (Vd), and clearance (Cl).

Hemostatic efficacy of the investigational product will be assessed by means of rotational thromboelastometry (ROTEM) measure of maximum clot firmness (MCF) at baseline and 1 hour post-infusion. Other thromboelastographic measures as well as standard coagulation tests will be also determined pre- and post-infusion.

Clinical safety, viral safety, and immunogenicity will be assessed in this clinical trial. Safety variables include adverse events (AEs), vital signs, physical assessments, laboratory tests, viral markers, and antibodies against human fibrinogen.

A monitoring plan will be implemented by the sponsor to carefully monitor and evaluate allergic/hypersensitivity reactions and thrombotic events during the study.

Stopping criteria have been established for immunogenic and thrombogenic events. If a single case of any these events is reported after a participants has been dosed with study drug, any further enrollment and dosing of participants in the study will be suspended until the event can be adequately assessed by the sponsor. The enrollment and dosing will only resume if the sponsor deems it is safe to do so.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants less than 70 years old.
2. Sign the written Informed Consent Form (ICF), or the subjects parent or legal guardian signs the ICF where applicable, and the subjects. Authorization Form where applicable. Pediatric subjects, as defined by local regulations, will be asked to sign an age appropriate assent form.
3. Subjects diagnosed with congenital fibrinogen deficiency manifested as afibrinogenemia.
4. Subjects with a fibrinogen level undetectable or equal or less than 30 mg/dL determined by both Clauss and antigen methods at baseline (sample drawn within 24 hours prior to infusion on Day 0 Visit) or at Screening Visit (sample drawn at least 14 days prior to infusion on Day 0 Visit).
5. Female subjects of child-bearing potential must have a negative test for pregnancy blood or urine human chorionic gonadotropin (HCG-based assay) at baseline (sample drawn within 24 hours prior to infusion on Day 0 Visit).
6. Female subjects of child-bearing potential and their partners have agreed to practice contraception using a method of proven reliability (i.e., hormonal methods; barrier methods; intrauterine devices methods) to prevent a pregnancy during the course of the clinical trial.
7. Subjects ants must be willing to comply with all aspects of the clinical trial protocol, including blood sampling, for the whole duration of the study.

Exclusion Criteria:

1. Subjects who received any fibrinogen-containing product within 21 days prior to Day 0 Visit - infusion day.
2. Subjects who present with active bleeding within 10 days prior to infusion on Day 0 Visit.
3. Subjects with acquired (secondary) fibrinogen deficiency.
4. Subjects diagnosed with dysfibrinogenemia.
5. Subjects with documented history of deep vein thrombosis, pulmonary embolism, or arterial thrombosis within 1 year prior to enrollment in this clinical trial.
6. Subjects with known antibodies against fibrinogen.
7. Subjects with a history of anaphylactic reactions or severe reactions to any blood-derived product.
8. Subjects with a history of intolerance to any component of the investigational products.
9. Subjects with a documented history of Immunoglobulin A (IgA) deficiency and antibodies against IgA.
10. Females who are pregnant or are breastfeeding.
11. Subjects with renal impairment (i.e., serum creatinine exceeds more than 2.0 times the upper limit of normal [ULN] at baseline [sample drawn within 24 hours prior to infusion on Day 0 Visit]).
12. Subjects with aspartate aminotransferase or alanine aminotransferase levels exceeding more than 2.5 times the ULN at baseline (sample drawn within 24 hours prior to infusion on Day 0 Visit).
13. Subjects with a history of chronic alcoholism or illicit drug addiction in the preceding 12 months prior to enrollment in this clinical trial.
14. Subjects with any medical condition which is likely to interfere with the evaluation of the study drugs and/or the satisfactory conduct of the clinical trial according to the investigator's judgment (e.g., congenital or acquired bleeding disorders other than congenital fibrinogen deficiency, planned surgery needing blood transfusion).
15. Subjects received aspirin-containing products and nonsteroidal anti-inflammatory drugs within 7 days prior to Day 0 Visit.
16. Subjects currently receiving, or having received within 3 months prior to enrollment into this clinical trial, any investigational drug or device.
17. Subjects who were previously administered the investigational product FIB Grifols during this clinical trial (i.e., every subject can only participate in the study once).
18. Subjects who are unlikely to adhere the protocol requirements, or are likely to be uncooperative, or unable to provide a storage serum sample prior to investigational drug infusion.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flora Peyvandi, MD, Study Chair — Centro Emofilia & Trombosi Angelo Bianchi Bonomi
Locations (6):
- Northshore Long Island Jewish Medical Center, New Hyde Park, New York, United States
- India (3):
  - S.S. Institute of Medical Sciences and Research Centre, Davangere, Karnataka
  - St. Johns Medical College and Hospital, Bangalore
  - Sahyadri Specialty Hospital, Pune
- Agenzia per l'Emofilia Centro di Riferimento Regionale per le Coaugulopatie Congenite A.O. di Carreggi, Florence, Italy
- Hôtel-Dieu de France Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in India, Lebanon, and the United States of America (USA) between 22 Jul 2016 (first participants first visit) and 11 Nov 2019 (last participant last visit).
Pre-assignment Details: A total of 26 participants were screened, out of which 24 participants were enrolled, of them 2 participants withdrew the consent prior to receiving the study treatment, and the remaining 22 participants received the study treatment.
Groups:
- FIB Grifols 70 mg/kg Body Weight: Participants received a single dose of slow intravenous infusion of Human Plasma-Derived Fibrinogen Concentrate Grifols (FIB Grifols) 70 milligram per kilogram (mg/kg) body weight, at a rate not exceeding 5 milliliter per minute (mL/min), on Day 0.
Period: Overall Study
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received infusion (at any dose) of the investigational product.
Groups:
- FIB Grifols 70 mg/kg Body Weight: Participants received a single dose of slow intravenous infusion of Human Plasma-Derived Fibrinogen Concentrate Grifols (FIB Grifols) 70 mg/kg body weight, at a rate not exceeding 5 mL/minute, on Day 0.
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.65 (9.523)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 22
  Asian | 14
  White | 8

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Fibrinogen Concentration-time Curve (AUC) From Time Zero to 14 Days (AUC0-14days) of FIB Grifols Determined by Clauss Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: AUC(0-14days) was calculated by a combination of linear and logarithmic trapezoidal methods and expressed in the unit of concentration × time. The linear trapezoidal method used for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method used for those arising from decreasing concentrations. Plasma fibrinogen activity determined by the Clauss method in the central laboratory of the study. Pharmacokinetic (PK) parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: The PK analysis population included all participants who had received study medication and had sufficient fibrinogen plasma concentration data to facilitate calculation of pharmacokinetic parameters. Here 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hour*grams per liter (h*g/L)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 10
hour*grams per liter (h*g/L) | 145.67 (43.441)

2. Primary Outcome: Area Under the Plasma Fibrinogen Concentration-time Curve (AUC) From Time Zero to 14 Days (AUC0-14days) of FIB Grifols Determined by Enzyme-Linked Immunosorbent Assay (ELISA) Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: AUC(0-14days) was calculated by a combination of linear and logarithmic trapezoidal methods and expressed in the unit of concentration × time. The linear trapezoidal method was used for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method was used for those arising from decreasing concentrations. Plasma fibrinogen activity was determined by the ELISA method in the central laboratory of the study. PK parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour*milligram per milliliter (h*mg/mL)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 10
hour*milligram per milliliter (h*mg/mL) | 186.63 (95.734)

3. Primary Outcome: AUC From Time Zero to Infinite Time (AUC0-infinity) of FIB Grifols Determined by Clauss Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: AUC0-infinity was calculated as AUC0-t + Ct/Kel, where (AUC0-t) was the area under the concentration versus (vs) time curve from time 0 to the time of last quantifiable concentration (Ct), and Kel was the apparent terminal first-order elimination rate constant, determined by linear regression analysis of the natural log-linear segment of the plasma concentration-time curve, expressed in time^-1 units (1/h). Plasma fibrinogen activity was determined by the Clauss method in the central laboratory of the study. PK parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*gram per liter (h*g/L)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 10
hours*gram per liter (h*g/L) | 166.78 (54.081)

4. Primary Outcome: AUC From Time Zero to Infinite Time (AUC0-infinity) of FIB Grifols Determined by ELISA Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: AUC0-infinity was calculated as AUC0-t + Ct/Kel, where (AUC0-t) was the area under the concentration vs. time curve from time 0 to the time of last quantifiable concentration (Ct), and Kel was the apparent terminal first-order elimination rate constant, determined by linear regression analysis of the natural log-linear segment of the plasma concentration-time curve, expressed in time^-1 units (1/h). Plasma fibrinogen activity was determined by the ELISA method in the central laboratory of the study. PK parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*mg/mL
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 7
h*mg/mL | 242.94 (117.567)

5. Primary Outcome: Maximum Observed Peak Plasma Fibrinogen Concentration (Cmax) of FIB Grifols Determined by Clauss Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: Cmax was obtained directly from the experimental data without interpolation. Plasma fibrinogen activity was determined by the Clauss method in the central laboratory of the study. PK parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 10
gram per liter (g/L) | 1.99 (0.404)

6. Primary Outcome: Maximum Observed Peak Plasma Fibrinogen Concentration (Cmax) of FIB Grifols Determined by ELISA Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: Cmax was obtained directly from directly from the experimental data without interpolation. Plasma fibrinogen activity was determined by the ELISA method in the central laboratory of the study. PK parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: The PK analysis population included all participants who had received study medication and had sufficient fibrinogen plasma concentration data to facilitate calculation of pharmacokinetic parameters. Here 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligram per milliliter (mg/mL)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 10
milligram per milliliter (mg/mL) | 2.88 (0.859)

7. Primary Outcome: Time to Reach Maximum Plasma Fibrinogen Concentration (Tmax) of FIB Grifols Determined by Clauss Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: Tmax was obtained directly from the experimental data without interpolation, expressed in time units (hour). Plasma fibrinogen activity was determined by the Clauss method in the central laboratory of the study.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: The PK analysis population included all participants who had received study medication and had sufficient fibrinogen plasma concentration data to facilitate calculation of pharmacokinetic parameters. Here, the 'number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 21
hour (h) | 1.40 [1.0 to 24.5]

8. Primary Outcome: Time to Reach Maximum Plasma Fibrinogen Concentration (Tmax) of FIB Grifols Determined by ELISA Method
Description: Tmax was obtained directly from the experimental data without interpolation, expressed in time units (hour). Plasma fibrinogen activity was determined by the ELISA method in the central laboratory of the study.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 7
Measure: Median (Full Range); unit: hour (h)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 21
hour (h) | 1.80 [1.1 to 24.5]

9. Primary Outcome: Apparent Terminal Half-life (t1/2) of FIB Grifols Determined by Clauss Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: t1/2 was the time measured for the concentration to decrease by one half. t1/2 calculated by natural log 2 divided by Kel and expressed in time units (hour). PK parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 10
hour (h) | 76.94 (20.215)

10. Primary Outcome: Apparent Terminal Half-life (t1/2) of FIB Grifols Determined by ELISA Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: as for outcome 9
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 7
hour (h) | 66.92 (16.789)

11. Primary Outcome: Mean Residence Time (MRT) of FIB Grifols Determined by Clauss Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: MRT was calculated by AUC0-inf/AUC0-inf - (T1/2), where AUC0-inf was the area under the first moment of the concentration vs. time curve from time 0 extrapolated to infinite time and T1/2 was the apparent terminal half-life of infusion. PK parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 10
hour (h) | 72.67 (12.185)

12. Primary Outcome: Mean Residence Time (MRT) of FIB Grifols Assessed Determined by ELISA Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: MRT was calculated by AUC0-inf/AUC0-inf - (T1/2), where AUC0-inf was the area under the first moment of the concentration vs. time curve from time 0 extrapolated to infinite time and T1/2 was the apparent terminal half life of infusion.PK parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 10
hour (h) | 62.64 (19.142)

13. Primary Outcome: Volume of Distribution (Vd) of FIB Grifols Determined by Clauss Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. PK parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 10
milliliter per kilogram (mL/kg) | 47.932 (7.5997)

14. Primary Outcome: Volume of Distribution (Vd) of FIB Grifols Determined by ELISA Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: as for outcome 13
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 7
mL/kg | 31.264 (10.9702)

15. Primary Outcome: Clearance (Cl) of FIB Grifols Determined By Clauss Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: Clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. PK parameters adjusted for baseline fibrinogen level calculated by deducting the pre-infusion fibrinogen concentration from the post-infusion concentrations before the calculation.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL per hour per kilogram (mL/h/kg)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 10
mL per hour per kilogram (mL/h/kg) | 0.454 (0.1216)

16. Primary Outcome: Clearance (Cl) of FIB Grifols Determined By ELISA Method, Dose Normalized to 70 mg/kg and Corrected for Baseline Concentration
Description: as for outcome 15
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 7
mL/h/kg | 0.341 (0.1360)

17. Primary Outcome: In Vivo Recovery (IVR) of FIB Grifols Determined by Clauss Method
Description: Incremental IVR was calculated for fibrinogen levels from the peak level recorded within and included the first four hours after the end of infusion and reported as milligram per deciliter per milligram per kilogram [mg/dL]/[mg/kg]. IVR was determined for every participants using the following formula: ([FIB max (mg/dL)] - [FIB pre-infusion (mg/dL)])/FIB administered (mg)/Body weight (kg), where the FIB max is the peak FIB activity within the first four hours after the end of infusion and FIB pre-infusion was the baseline FIB activity level of the participant. FIB administered was the actual administered dose calculated using the actual volume administered to the participant, the declared potency, and the true concentration of FIB in the batch used.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)/ (mg/kg)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 21
milligram per deciliter (mg/dL)/ (mg/kg) | 2.380 (0.6689)

18. Primary Outcome: In Vivo Recovery (IVR) of FIB Grifols Determined by ELISA Method
Description: Incremental IVR was calculated for fibrinogen levels from the peak level recorded within and included the first four hours after the end of infusion and reported as milligram per deciliter per milligram per kilogram [mg/dL]/[mg/kg]. IVR was determined for every participants using the following formula: ([FIB max (mg/dL)] - [FIB pre-infusion (mg/dL)])/FIB administered (mg)/Body weight (kg), where the FIB max is the peak FIB activity within the first four hours after the end of infusion and FIB pre-infusion was the baseline FIB activity level of the participants. FIB administered was the actual administered dose calculated using the actual volume administered to the participants, the declared potency, and the true concentration of FIB in the batch used.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216 and 336 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (mg/dL)/(mg/kg)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 21
(mg/dL)/(mg/kg) | 3.474 (1.3607)

19. Primary Outcome: Mean Change on Maximum Clot Firmness (MCF) From Baseline to 1-hour Post-infusion
Description: MCF was as a functional parameter of blood's ability to coagulate, provides an indirect measure of hemostatic efficacy of replacement treatment with fibrinogen concentrates in participants with fibrinogen deficiency. Rotational thromboelastography (ROTEM) was performed on frozen plasma samples by the central laboratory to measure MCF. Undetectable MCF values were set to 0.
Time Frame: Baseline to 1-hour post-infusion
Population: The Evaluable population included all participants who received Investigational Product (IP) at any amount and who had at least two measurements, pre-infusion MCF and 1-hour post-infusion MCF measurements by ROTEM. Here 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 21
millimeter (mm) | 10.71 (4.122)

20. Secondary Outcome: Mean Change in Clotting Time (CT) From Baseline to 1-hour Post-infusion
Description: Difference in adult participants plasma samples in CT from baseline to 1-hour post-infusion indicated the hemostatic efficacy of the treatment with fibrinogen concentrate in participants with fibrinogen deficiency.
Time Frame: Baseline to 1-hour post-infusion
Population: The Evaluable population included participants who received investigational product at any amount and who had at least 2 measurements pre-infusion MCF and 1-hour post-infusion MCF measurements by ROTEM. Here 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Seconds (sec)
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 1
Seconds (sec) | -3462.0 (NA) — Standard deviation could not be estimated as there was only 1 participant with detectable baseline CT value and thus analyzed, undetectable CT values were set to missing.

21. Secondary Outcome: Clot Formation Time (CFT) at 1-hour Post-infusion
Description: CFT value in participants plasma samples in CFT at 1-hour post-infusion indicated the hemostatic efficacy of the treatment with fibrinogen concentrate in participants with fibrinogen deficiency.
Time Frame: 1-hour post-infusion
Population: Evaluable population included participants who received investigational product at any amount and who had at least 2 measurements pre-infusion MCF and 1-hour post-infusion MCF measurements by ROTEM. Here 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 1
sec | 68.0 (NA) — Standard deviation could not be estimated as there was only 1 participant with detectable baseline CFT value and thus analyzed, undetectable CFT values were set to missing.

22. Secondary Outcome: Mean Change in Alpha Angle (α) From Baseline to 1-hour Post-infusion
Description: Difference in participants plasma samples in alpha angle from baseline to 1-hour post-infusion indicated the hemostatic efficacy of the treatment with fibrinogen concentrate in participants with fibrinogen deficiency.
Time Frame: Baseline to 1-hour post-infusion
Population: The Evaluable population included all participants who received at any amount and who had at least two measurements, pre-infusion MCF and 1-hour post-infusion MCF measurements by ROTEM. Here 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 21
degree | 34.9 (34.52)

23. Secondary Outcome: Mean Change in Prothrombin Time (PT) From Baseline to 1-hour Post-infusion
Description: Difference in the participants plasma samples standard coagulation tests from baseline to 1-hour post-infusion indicated hemostatic efficacy of the treatment with fibrinogen concentrate in participants with fibrinogen deficiency.
Time Frame: Baseline to 1-hour post-infusion
Population: The Evaluable population included all participants who received at any amount and who had at least two measurements, pre-infusion MCF and 1-hour post-infusion MCF measurements by ROTEM. Here 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 17
sec | -102.79 (2.101)

24. Secondary Outcome: Mean Change in Thrombin Time (TT) From Baseline to 1-hour Post-infusion
Description: as for outcome 23
Time Frame: Baseline to 1-hour post-infusion
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 19
sec | -200.41 (58.178)

25. Secondary Outcome: Mean Change in Activated Partial Thromboplastin Time (aPTT) From Baseline to 1-hour Post-infusion
Description: Difference in participants plasma samples standard coagulation tests from baseline to 1-hour post-infusion indicated hemostatic efficacy of the treatment with a fibrinogen concentrate in participants with fibrinogen deficiency.
Time Frame: Baseline to 1-hour post-infusion
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 19
sec | -97.16 (10.580)

26. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study drug which may or may not have a causal relationship with the study drug. SAE was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-participants hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Treatment-emergent defined as adverse events/serious adverse events that started or worsened on or after the start of the investigational product infusion.
Time Frame: From the start of the investigation product infusion up to Week 4
Population: The Safety population included all participants who received infusion (at any dose) of the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | FIB Grifols 70 mg/kg Body Weight
Number analyzed (Participants) | 22
Participants
  Participants with AEs | 9
  Participants with Serious AEs | 0

ADVERSE EVENTS:
Time Frame: From the start of the investigational product infusion up to Week 4
Description: The Safety population included all participants who received infusion (at any dose) of the IP.
Groups:
- FIB Grifols 70 mg/kg Body Weight: Participants received a single dose of slow IV infusion of FIB Grifols 70 mg/kg body weight, at a rate not exceeding 5 mL/minute, on Day 0.
Arm/Group | FIB Grifols 70 mg/kg Body Weight
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 9/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FIB Grifols 70 mg/kg Body Weight (N=22)
Abdominal pain (Gastrointestinal disorders) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Blood pressure diastolic decreased (Investigations) | 1
Blood pressure systolic decreased (Investigations) | 1
Body temperature increased (Investigations) | 1
Heart rate increased (Investigations) | 1
Headache (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT02281500/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT02281500/SAP_001.pdf